CLINICAL TRIAL: NCT05979350
Title: Impact of Incorporating Metagenomic Next-generation Sequencing in the Management of Pneumonia on Diagnostic Efficiency and Outcomes: A Randomized Controlled Trial
Brief Title: Metagenomic NGS for Diagnosis of Pneumonia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital Hsin-Chu Branch (Other); Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202305104RINB
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Pneumonia; Diagnosis
Keywords: diagnosis; next-generation sequencing; outcome; pneumonia
MeSH Terms: conditions — Pneumonia; Disease

STUDY DESIGN:
Intervention Model Description: Paralleled 1:1 randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care group (Active Comparator): Endotracheal aspirates, blood samples, urine samples, and nasopharyngeal swabs were obtained from the patients as soon as possible after ICU admission. Bacterial culture was performed, with the use of standard techniques, on blood samples and endotracheal aspirates. Urine antigen detection was performed for detection of L. pneumophila and S. pneumoniae. A PCR assay was performed on nasopharyngeal swabs for the detection of influenza A and B viruses and SARS-CoV-2 viruses. Fungal or mycobacterial detections, and whether to use multiplex PCR for pathogen detection, such as the FilmArray system, were determined at the discretion of the physicians.
  Interventions: Diagnostic Test: Standard work-up for pneumonia
- mNGS group (Experimental): Subjects assigned to the mNGS group will receive etiology work-up followed the protocol used in the standard care group and additional mNGS testing for two specimen of mini-bronchoalveolar lavage and one specimen of blood samples retrieved at the same time of standard work-up.
  Interventions: Diagnostic Test: Metagenomic next-generation sequencing

INTERVENTIONS:
Diagnostic Test: Metagenomic next-generation sequencing — Metagenomic NGS testing for pathogen identification will be done for airway and blood specimens using APGseq ® (Asia Pathogenomics, New Taipei City, Taiwan). The sample preparation for mNGS testing was as follows: 5-10 mL of whole blood were centrifuged at 1,600g for 10 min at 4°C to separate the plasma. Plasma samples were transferred to 2 mL sterile tubes for the following DNA or RNA extraction. In general, 300ul of plasma sample was used for DNA extraction. Total genomic DNA from samples were extracted using the column-based method (e.g. QIAamp DNA Microbiome Kit, Qiagen for DNA extraction; or QIAamp Viral RNA Mini Kit, Qiagen for RNA extraction, respectively), following the manufacturer's operational manual. The RNA was reverse transcribed and synthesized to double-stranded complementary DNA (ds cDNA) with SuperScript II Reverse Transcription Kit (Invitrogen).
  Arms: mNGS group
Diagnostic Test: Standard work-up for pneumonia — Endotracheal aspirates, blood samples, urine samples, and nasopharyngeal swabs were obtained from the patients as soon as possible after ICU admission. Bacterial culture was performed, with the use of standard techniques, on blood samples and endotracheal aspirates. Urine antigen detection was performed for detection of L. pneumophila and S. pneumoniae. A PCR assay was performed on nasopharyngeal swabs for the detection of influenza A and B viruses and SARS-CoV-2 viruses. Fungal or mycobacterial detections, and whether to use multiplex PCR for pathogen detection, such as the FilmArray system, were determined at the discretion of the physicians.
  Arms: Standard care group

SUMMARY:
In this randomized controlled trial, we aim to evaluate the efficacy of incorporating mNGS in the management of pneumonia on efficiency and accuracy of causative pathogen identification, proportion of participants with effective antimicrobial therapy, length of hospitalization, and mortality.

DETAILED DESCRIPTION:
This is an open-label, randomized, multi-center, phase 2 study that will evaluate the efficacy of incorporating mNGS in the management of severe pneumonia on accuracy and efficiency of achieving definite diagnosis of identifying causative pathogens of pneumonia, appropriate antimicrobial therapy and patient outcomes. The diagnosis of pneumonia requires radiological evidence of pneumonia and at least two of the following clinical criteria: new, or worsening cough, new or worsening expectoration of sputum, new or worsening dyspnea, hemoptysis, pleuritic chest pain, and fever (≥38.0°C). Severe pneumonia is defined as pneumonia with hypoxemia requiring orotracheal intubation and mechanical ventilation support.

Written informed consent is needed from the eligible subjects or from their legal guardian at the time of recruitment. After completing informed consent, subjects will be randomized with a 1:1 allocation ratio via a web-based randomization system to receive standard of care (SOC) using culture and serology based work-up for pathogen detection or SOC with additional mNGS method using APGseq ® (Asia Pathogenomics, New Taipei City, Taiwan) for pathogen detection. The treatment for pneumonia is suggested following the Taiwan Guidelines for the Management of Pneumonia published in 2018. After randomization, the subjects will be followed until death, discharged from the hospital or 28 days after randomization whichever comes first. The total study duration is expected to be two years from the first subject enrolled to the final analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Presenting to the ICU with a diagnosis of pneumonia (fulfilled with both radiographic and clinical criteria)
2. Adults aged ≥18 years
3. Orotracheally intubated
4. ICU admission for <24 hours
5. APACHE II score <35 on ICU admission

Exclusion Criteria:

1. Life expectancy below 4 weeks
2. With an existing directive to withhold life-sustaining treatment
3. Patients not willing or able to provide a lower respiratory tract sample at ICU admission
4. Previous work-up has identified specific pathogens which can account for the index event of pneumonia
5. Multiplex PCR or NGS testing has been done for pathogen detection before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Time to achieving definite diagnosis in modified intention-to-treat (mITT) analysis. | 7 days
  Cumulative probability of achieving definite diagnosis in terms of accurately identifying causative pathogens of pneumonia, estimated by the Kaplan-Meier method in a time frame of 7 days in modified intention-to-treat (mITT) analysis.

SECONDARY OUTCOMES:
Time to achieving definite diagnosis in intention-to-treat analysis. | 7 days
  To test the robustness of mITT analysis for the primary study endpoint as compared with standard ITT analysis. (Sensitivity analysis)
Pathogen detection rate between two groups by the 72th hour. | 72 hours
  Proportion of participants with accurate diagnosis for the causative pathogens of pneumonia by the 72th hour after randomization in mITT analysis.
Pathogen detection rate between two groups by the end of study. | 28 days
  Proportion of participants with accurate diagnosis for the causative pathogens of pneumonia by the day 28 after randomization in mITT analysis.
Impact of mNGS on appropriate antibiotic prescription. | 72 hours
  Proportion of participants on effective antimicrobial therapy by the 72th hour after randomization in mITT analysis.
28-day mortality in mITT analysis. | 28 days
  Kaplan-Meier curves of 28-day survival using mITT cohort. Log-rank tests are used to test statistical significance.
28-day mortality in ITT analysis (total cohort). | 28 days
  Kaplan-Meier curves of 28-day survival using total cohort. Log-rank tests are used to test statistical significance.
Impact of mNGS on respiratory and mortality outcome. | 28 days
  Ventilator-free days in 28 days using the mITT cohort. Wilcoxon rank-sum test is used to test statistical significance.
Impact of mNGS on the length of ICU stay | ICU discharge or 28 days
  Curves of alive ICU discharge in 28 days after randomization using the Fine-Gray model. Death will treated as a competing risk.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Yuan Ruan, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No